CLINICAL TRIAL: NCT06842641
Title: A Cluster Randomized Controlled Trial (cRCT) Evaluating the Effects of Cool Roofs on Health Outcomes Using Smartwatches in Ouagadougou, Burkina Faso
Brief Title: Assessing the Effect of Cool Roofs on Health Using Smartwatches in Ouagadougou, Burkina Faso
Acronym: REFLECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Supérieur des Sciences de la Population (Other)
Collaborators: University of Auckland, New Zealand (Other); Heidelberg University (Other); London School of Hygiene and Tropical Medicine (Other); Rutgers University (Other); Boston University (Other); Secretaría de Educación Pública, México (Other Government); University of Ouagadougou, Burkina Faso (Other); Indian Institute of Public Health, India (Other); The Tindall Foundation (Other); Habitat for Humanity (Other); Pacific Community (Other); Labfront (Industry); Cognifit (Unknown); Resene (Industry); SOPREMA (Unknown); EPS (Unknown); Sika (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3728163; 226745/Z/22/Z (Other: Wellcome Trust UK)
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Heart Rate; All-day Steps; Distance Walked; Active Minutes; Moderate-intensity Activity Minutes; Sleep Quantity; Time in Sleep Stages; Awake Duration; Sleep Score
Keywords: Hot Temperature; Humidity; Housing; Wearable; Smartwatch; Heart rate; Cardiovascular; Physical activity; Sleep; Cool roof
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Trial participants will be aware of the intervention to which they have been allocated, and the research fieldworkers will be aware of the intervention allocation. The trial steering committee members and trial statistician will remain blinded until the end of trial period and data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Households will receive sunlight reflecting 'cool roof' coating on their roofs.
  Interventions: Other: Cool roof
- Control (No Intervention): No cool roof application. Households will keep their original roofing for the duration of the trial.

INTERVENTIONS:
Other: Cool roof — Cool roofs are a sunlight reflecting roof coating that can reduce indoor temperature. Cool roofs have high solar reflectance (reflecting the ultraviolet and visible wavelengths of sunlight, reducing heat transfer to the surface of a roof) and high thermal emittance (radiating absorbed solar energy
  Arms: Intervention

SUMMARY:
Ambient air temperatures in Africa, have broken record highs in 2024. Solutions are needed to build heat resilience in communities and adapt to increasing heat from climate change. Sunlight-reflecting cool roof coatings may passively reduce indoor temperatures and energy use to protect home occupants from extreme heat. Occupants living in poor housing conditions- for example in informal settlements, slums, and low-socioeconomic households - are susceptible to increased heat exposure.

Heat exposure can instigate and worsen numerous physical, mental and social health conditions. The worst adverse health effects are experienced in communities that are least able to adapt to heat exposure. By reducing indoor temperatures, cool roof application may improve heart health, sleep and physical activity in household occupants.

The long-term research goal is to identify viable passive housing adaptation technologies with proven health benefits to reduce the burden of heat stress in communities affected by heat. To meet this goal, the investigators will use smartwatches to measure the effects cool roof application on heart health, sleep and physical activity in Ouagadougou, Burkina Faso.

DETAILED DESCRIPTION:
Increasing heat exposure from climate change is causing and exacerbating heat-related illnesses in millions worldwide - particularly in low resource settings. June 2024 was the 13th consecutive hottest month on record globally - shattering previous records. Heat exposure can instigate and worsen numerous health conditions. Adaptation is essential for protecting people from increasing heat exposure. The built environment, especially homes, are ideal for deploying interventions to reduce heat exposure and accelerate adaptation efforts. However, evidence is currently lacking on a global scale - generated through empirical studies - guiding the uptake of interventions to reduce indoor heat stress in low resource settings.

Sunlight-reflecting cool roof coatings passively reduce indoor temperatures and lower energy use, offering protection to home occupants from extreme heat. Continuous monitoring of health and wellbeing using smartwatches can provide insight into important parameters such as heart rate, sleep and physical activity - which are all affected by heat. Using smartwatches, the investigators will also continuously measure health and wellbeing outcomes during the day and night. The investigators will conduct a study to investigate the effects of cool-roof use on heart rate, sleep and physical activity in Ouagadougou, Burkina Faso (sub-Saharan Africa, where people experience a triple burden from heat exposure, chronic health issues and vulnerable housing conditions (slums, informal settlements and low socioeconomic housing).

This trial will quantify whether cool roofs are an effective passive home cooling intervention with beneficial health effects for vulnerable populations in Burkina Faso. Findings will inform global policy responses on scaling cool roof implementation to protect people from increasing heat exposure driven by climate change.

ELIGIBILITY:
Inclusion Criteria:

* • Permanent household resident

Exclusion Criteria:

* • Roof damage, inaccessible or instability of roof adversely affecting cool roof coating application.

  * Participant unable to provide written/verbal informed consent. Participants will be excluded if they are not willing or able to wear a smartwatch.
  * One participant per household.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Heart rate | The outcome will be measured at 15-second intervals continuously throughout each 12-month period, with participants wearing the device for at least two weeks per month to capture consistent data points.
  Heart rate in beats per minute measured at 15-second intervals using Garmin Vivosmart 5 devices. Measurements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.

SECONDARY OUTCOMES:
All-day steps | Measurements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The number of steps measured daily using Garmin Vivosmart 5 devices.
Distance walked | Measurements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The total distance walked daily using Garmin Vivosmart 5 devices
Active minutes | Measurements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The total number of minutes of active exercise daily using Garmin Vivosmart 5 devices.
Moderate-intensity activity minutes | Measurements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The total number of minutes of moderate-intensity activity daily using Garmin Vivosmart 5 devices.
Vigorous-intensity activity duration | Measurements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The total number of minutes of vigorous-intensity activity daily using Garmin Vivosmart 5 devices.
Sleep quantity | Measurements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The number of hours spent asleep each night using Garmin Vivosmart 5 devices.
Time in sleep stages | Measurements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The number of hours spent in sleep stages each night using Garmin Vivosmart 5 devices.
Awake duration | Measurements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The number of hours spent awake during sleep time each night using Garmin Vivosmart 5 devices.
Sleep score | Measurements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The Garmin sleep score (0-100) each night using Garmin Vivosmart 5 devices.

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Bunker, Doctor of Phylosophy (Ph.D), Principal Investigator — Heidelberg University
Locations (1):
- Ouagadougou Health and Demographic Surveillance System, Ouagadougou, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Data that can be shared unconditionally underpinning the published research articles will be made available to other researchers at the time of publication, and data will be linked via the article DOI. Data that cannot be unconditionally shared upon publication owing to confidentiality or data protection requirements will be identified as such and a contact email will be provided in relevant publications for data access enquiries by other researchers. Individual names of study participants and identifying factors will be removed prior to data sharing.
  It is expected that demographic data of people at the study sites (family size and composition, basic socioeconomic indicators) may contain personally identifiable information and location data. All such data will be removed prior to storage on online data repositories and therefore will be available to be publicly shared at the time of publication of manuscripts.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the time of publication.